CLINICAL TRIAL: NCT03538132
Title: Patients' Perception on Bone Biomaterials Used in Dentistry : a Multicentric Study
Brief Title: Patients' Perception on Bone Grafts
Acronym: PEPABIO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0456
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Dental Treatment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dental regenerative techniques — dental regenerative techniques

SUMMARY:
The goal of this study is to collect the patients' opinion about the different types of bone graft, to assess which are the most rejected by the patients and if the demographic variables (such as the gender or the age) and the level of education influence their decision.

DETAILED DESCRIPTION:
Nowadays, many procedures may need regenerative techniques. Some studies have already assessed the patients' opinion regarding soft tissue grafts, some investigators have centered their studies on the techniques' efficiency without assessing the patient's perception.

In addition to grafts harvested from the patient himself (autologous graft), bone graft can also be obtained from animals (xenograft), human cadavers (allograft) and synthetic materials (alloplastic graft). Patients may have ethical, religious or medical concerns about the origin of each bone graft, which could lead them to reject the use of certain types of bone graft in their surgery.

The aim of this multicenter study, which surveys patients from five university clinics in Portugal, Italy, Spain, France and Chile, is to analyze patients' opinions regarding the source of bone grafts.

A survey composed of 10 questions is submitted to the patients. They are asked about the degree of acceptance/rejection of each graft and their reasons for rejecting it.

In France, the survey will be presented to 100 patients having dental treatments in the "Centre de Soins Dentaires" of Montpellier from december of 2017 to june of 2018.

Eligibility criterias : adult (18 years of age or older), able to read and write in the local language, not under the influence of alcohol or drugs, had not previously undergone any surgery involving bone graft or bone augmentation, able to understand and follow the indications for the survey completion, willingness to participate in the study

Data obtained :

The survey is formed by two parts. The first part records the participant's demographic data, such as: gender, age, education level and religion: participants are asked, "Do you profess a religious faith?" (yes/no). In case of a positive answer, they are asked to which religion they adhere.

The second part of the survey consists of 10 questions regarding acceptance/rejection of the bone grafts. Patients are asked to mark only one answer, which best aligned with their opinion.

Questions are classified as follows:

Five closed-ended questions (with lists of possible answers) about the level of acceptance of each type of bone graft (acceptance, conditional acceptance or refusal).

Three open-ended questions (i.e., the patients' spontaneous answers were recorded).

Two mixed questions that aimed to identify the reasons for refusal (if applicable).

ELIGIBILITY:
Inclusion criteria:

* Adult (18 years old or more)
* Able to read and write
* Not under the influence of alcohol or drugs
* Had not previously undergone any surgery involving bone graft or bone augmentation.

Exclusion criteria:

- Any patient who doesn't fullfill the inclusion criterias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that had been treated in the "Centre de soins, d'enseignements et de recherches dentaires de l'Université de Montpellier" between December of 2017 and June of 2018.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of patients' opinions on the different types of biomaterials used in regenerative techniques. | 1 day
  Evaluation of patients' opinions on the different types of biomaterials used in regenerative techniques through a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marie ORDONNEAU, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC